CLINICAL TRIAL: NCT05178524
Title: Clinical Study on BIFICO Accelerating Postoperative Liver Function Recovery in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang Bi Xiang, MD, Chairman of Department of General Surgery, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20210532
Record Dates: First submitted 2021-11-21; First posted 2022-01-05 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-05

CONDITIONS: Gut Microbiota; Hepatocellular Carcinoma; Bifidobacterium
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifico Group (Experimental): Continued administration during perioperative period
  Interventions: Drug: BIFICO
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Drug: BIFICO — Live combined Bifidobacterium, Lactobacillus and Enterococcus Capsules
  Arms: Bifico Group

SUMMARY:
On the basis of previous studies, this study intends to explore the effect of BIFICO on liver function recovery of patients with hepatocellular carcinoma (HCC) after surgery, so as to provide a new method for accelerating liver function recovery of HCC patients during perioperative period.

This project is an open, randomized, blank-controlled clinical study. Liver resection patients were randomly divided into two groups, one group received continuous administration of BIFICO during perioperative period, and the dosage was controlled according to the instructions. The other group was a blank control. Stool samples were collected at three time points (before medication, before and after surgery) in two groups. Statistical analysis was performed to compare the differences of postoperative liver function and preoperative and postoperative gut microbiota between the two groups.

Through this study, the investigators aimed to verify the beneficial changes of intestinal microflora in HCC patients with BIFICO during perioperative period .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors in the digestive system, with a high incidence in the world and the third highest mortality rate among all malignant tumors in China. In recent years, studies have found that intestinal microflora disorder can also promote the occurrence and development of HCC through various ways, such as endotoxemia, metabolic disorders, and increased risk of exposure to HBV and aflatoxin. In the treatment of HCC, in addition to the traditional comprehensive treatment based on surgical resection, the treatment for intestinal microflora disorder also plays a unique role in improving prognosis and alleviating complications.

At present, increasing the number of beneficial bacteria through probiotics is an important method to restore the ecological balance of intestinal microorganisms. Probiotics can maintain the balance of intestinal microecology and the integrity of intestinal mucosal barrier by inhibiting the growth of harmful bacteria, stimulating fermentation, stimulating the proliferation of intestinal mucosal cells and activating the immune system.

The preliminary study of this project has shown that the difference of intestinal flora in patients with HCC has a certain impact on the recovery speed of liver function after hepatectomy, and the core flora affecting postoperative liver function is bifidobacteria. Meanwhile, animal experiments have also verified that bifidobacteria can improve the postoperative liver function of mice. Therefore, improving the structure and environment of intestinal microorganisms, increasing the colonization of beneficial bacteria and enhancing the diversity of bacteria are very important to accelerate the recovery of liver function after hepatectomy for patients with HCC.

In this project, it is planned to use bifidobacteria-rich BIFICO as an intervention drug to sustained medication in the perioperative period of hepatectomy patients with HCC, and observe the recovery of postoperative liver function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 80 years old
* Imaging diagnosis of primary HCC, without other malignancies
* No antibiotic treatment within two weeks before surgery
* Regular diet and no severe diarrhea
* Laparoscopic or open hepatectomy is performed

Exclusion Criteria:

* No liver resection is performed
* No preoperative or postoperative stool samples during the perioperative period
* Pathological diagnosis is not HCC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of liver function recovery with total bilirubin and prothrombin activity | Five days after the surgery
  The liver function recovery of the two groups on the fifth day after surgery was compared, and t-test was used to verify whether there was a significant difference between the two groups. Total bilirubin and prothrombin activity were used to assess liver function.
The alpha and beta diversity analysis of gut microbiota | Baseline (Before the surgery)
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota between two groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
The alpha and beta diversity analysis of gut microbiota | Five days after the surgery
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota between two groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Species composition and differential analysis of gut microbiota | Baseline (Before the surgery)
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the community histogram, the community heatmap and the Wayne map will be used to analyze the species composition of the sample; the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition between the two groups. To further screen the species with significant differences, the LEfSe difference discriminant analysis will be used.
Species composition and differential analysis of gut microbiota | Five days after the surgery
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the community histogram, the community heatmap and the Wayne map will be used to analyze the species composition of the sample; the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition between the two groups. To further screen the species with significant differences, the LEfSe difference discriminant analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Bixiang Zhang, Study Chair — Tongji Hospital; Jingjing Yu, Principal Investigator — Tongji Hospital
Locations (1):
- The hepatic surgery of Tongji hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yu J, Zhu P, Shi L, Gao N, Li Y, Shu C, Xu Y, Yu Y, He J, Guo D, Zhang X, Wang X, Shao S, Dong W, Wang Y, Zhang W, Zhang W, Chen WH, Chen X, Liu Z, Yang X, Zhang B. Bifidobacterium longum promotes postoperative liver function recovery in patients with hepatocellular carcinoma. Cell Host Microbe. 2024 Jan 10;32(1):131-144.e6. doi: 10.1016/j.chom.2023.11.011. Epub 2023 Dec 12. PMID 38091982